CLINICAL TRIAL: NCT00788736
Title: Development and Validation of Clinical Prediction Rules for Bleeding for Patients on Anticoagulant Therapy for Venous Thromboembolism
Brief Title: Predicting Bleeding Risk on Anticoagulant Therapy for Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: OHREB 2008270-01H; MOP130388 (Other: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; long-term oral anticoagulant therapy; warfarin; bleeding risk; clinical prediction rule; predictors; deep vein thrombosis; pulmonary embolism; vitamin k antagonist; side effect
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects may consent to optional DNA and plasma banking
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of the study is to develop or validate a clinical prediction rule for major bleeding in patients on oral anticoagulant therapy who have been safely anticoagulated without bleeding or venous thromboembolism (VTE) recurrence for at least 3 months since diagnosis and are being considered for long-term oral anticoagulant therapy.

DETAILED DESCRIPTION:
Oral anticoagulant therapy for patients who are at risk of developing blood clotting problems is used by between 400,000-600,000 Canadians annually. The use of this drug represents the most common cause of patient adverse medical outcomes due to medical errors. Furthermore, many patients have adverse outcomes using these drugs because physicians are not able to predict which patients are likely to have bleeding outcomes. Much effort has gone into developing ways to predict which patients are at risk of clotting but almost no work has gone into ways of predicting which patients would be at high risk of bleeding. This information is required to balance off the risk-benefits and to enable physicians and patients to understand the risks and benefits of taking these medications. Our study will develop a tool that can be used to predict bleeding risk in patients taking oral anticoagulant therapy. It will enable more informed decision making by both physicians and patients and will result in better control of the use of these drugs. In addition, patients who are at risk for being difficult to accurately dose on oral anticoagulants will be identified through our study.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old
* provoked or unprovoked venous thromboembolism
* objectively confirmed venous thromboembolism
* treated with an oral anticoagulant(vitamin K antagonist or new oral anticoagulant) for at least 3 months with plans to continue long-term
* if taking a vitamin K antagonist; INR target is between 2.0-3.0
* if taking a vitamin K antagonist; must have taken it for the last 3 consecutive weeks (minimum)

Exclusion Criteria:

* major bleeding while taking oral anticoagulants
* active bleeding at study enrollment
* active cancer - current or at the time of VTE diagnosis
* unable to provide written informed consent
* refusal to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients being treated for venous thromboembolism
Sampling Method: Non-Probability Sample
Enrollment: 2537 (Actual)
Dates: Start 2008-09; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Major bleeding (International Society on Thrombosis and Haemostasis(ISTH) criteria) | ongoing for 3-7 years with follow-up phone calls at 6-month intervals

SECONDARY OUTCOMES:
Clinically relevant non-major bleeding (International Society on Thrombosis and Haemostasis(ISTH) criteria) | ongoing for 3-7 years with follow-up phone calls at 6-month intervals
recurrent venous thromboembolism | ongoing for 3-7 years with follow-up phone calls at 6-month intervals
death (all causes) | ongoing for 3-7 years with follow-up phone calls at 6-month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Phil S Wells, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (12):
- United States (2):
  - Lahey Clinic, Burlington, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
- Canada (9):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Sir Mortimer B Davis Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Centre, Montreal, Quebec
  - Hopital du Sacre Coeur de Montreal, Montreal, Quebec
- Oxford Haemophilia and Thrombosis Centre, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided